CLINICAL TRIAL: NCT02894489
Title: Changes of Visual Function, Ocular Surface Structures and Physiology After Long-Termed Contact Lens Wear
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, Hsiao Sang Chu, MD, Principal Investigator, National Taiwan University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201508075RINC
Record Dates: First submitted 2016-08-30; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Ocular Surface Disease; Keratoconus; Irregular Astigmatism
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- corneal lenses (Experimental): patients that wear corneal lenses ( Hiclear Rigid Gas Permeable Lenses)
  Interventions: Device: corneal lenses
- large diameter lenses (Experimental): patients that wear scleral lenses (Paragon Normaleyes)
  Interventions: Device: large diameter lenses

INTERVENTIONS:
Device: corneal lenses — wear corneal lenses on daily basis
  Arms: corneal lenses
Device: large diameter lenses
  Arms: large diameter lenses

SUMMARY:
Our study is aimed to observe the long termed effect of contact lens wear on ocular surface, especially focused on visual function and ocular inflammation mediators.

DETAILED DESCRIPTION:
Contact lens fitting are important treatments for many ocular diseases as they provide three main therapeutic applications: visual correction, protection of ocular surface, and cosmetic or sport purposes. The ophthalmology department of NTUH has set up contact lens special clinic as one of our comprehensive refractive services. The investigators provided corneal lenses or Rose K lenses for optical correction of keratoconus patients; the investigators also fitted large scleral lenses for the correction of irregular astigmatism for post-penetrating keratoplasty and post-refractive surgery patients. In addition, contact lenses can be an adjuvant therapy for ocular surface disorders as severe dry eye and limbal insufficiency. There were researches that proved the inflammatory mediators and neutrophils increased after long-termed wear of silicon hydrogel soft lenses or over night orthokeratology lenses. They also concluded that lens wear affected corneal epithelial proliferation. However, the physiological changes after long-termed wear of large diameter scleral lenses are still pending. In addition, we still do not understand the lens effects on high order aberration and ocular surface structures. The purpose of our study is to analyze the epidemiologic data and treatment results of the patients fitted with specialty lenses in our contact lens clinic from Aug 2016 to Aug 2018. Patients will be categorized into different groups by the diagnoses and the type of lens wear. After 6 months of follow up, the change of visual acuity, visual function related quality of life, the changes of ocular surface structures and physiology will be analyzed. The investigators hope to share the experiences of specialty contact lens fitting and understand the effects of long-term contact lens wear on ocular surface.

ELIGIBILITY:
Inclusion Criteria:

* age 20 to 65
* contact lens wear
* willing to be followed for at least 6 months

Exclusion Criteria:

* active ocular infection
* active corneal melting
* inability to follow lens cleaning instructions
* pregnancy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Ocular inflammatory mediators | 6 months
  to monitor the change of tear inflammatory mediators 6 months after lens wear

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao Sang Chu, MD, MS, Principal Investigator — Department of Ophthalmology, NTUH
Locations (1):
- Hsiao Sang Chu, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
for publication